CLINICAL TRIAL: NCT06924710
Title: A Prospective Multicenter Randomized Controlled Study of Adaptive Therapy in Resected Stage ⅠA2-Ⅱ NSCLC Patients With Undetectable MRD
Brief Title: Adaptive Therapy for Resected Stage ⅠA2-Ⅱ NSCLC Patients With Undetectable MRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Tianjin Chest Hospital (Other); Peking University First Hospital (Other); Bethune First Hospital of Jilin University (Unknown); Beijing Friendship Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Liaoning Cancer Hospital & Institute (Other); Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024KT205; ZLRK202524 (Other Grant/Funding Number: Beijing Hospitals Authority)
Record Dates: First submitted 2025-03-20; First posted 2025-04-11 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-04

CONDITIONS: NSCLC
Keywords: MRD; ctDNA
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Therapy (Active Comparator): Patients in this group will be treated following the guidelines.
  Interventions: Drug: Standard Therapy
- Adaptive Therapy (Experimental): Patients in this group will undergo closely MRD and imaging monitoring without adjuvant therapy if the MRD was negative.
  Interventions: Other: Adaptive Therapy

INTERVENTIONS:
Drug: Standard Therapy — For patients with negative EGFR/ALK mutation, adjuvant chemotherapy or adjuvant chemotherapy combined with immunotherapy was administered, for patients with positive EGFR/ALK mutation, targeted therapy was administered.
  Arms: Standard Therapy
Other: Adaptive Therapy — Patients will be under close MRD and imaging monitoring without adjuvant therapy if the MRD was negative.
  Arms: Adaptive Therapy

SUMMARY:
It is a prospective, multicenter, randomized controlled trial to investigate the predictive value of MRD on adjuvant therapy. Stage IA2-II resected NSCLC patients will undergo two-round MRD tests after surgery, first in 3-7 days and second in 1 month after surgery. And patients who confirm two-round landmark undetectable MRD will be enrolled and randomly assigned to the conventional treatment group or the adaptive therapy group . Patients in the the adaptive therapy group will undergo closely MRD and imaging monitoring without adjuvant therapy if the MRD was negative.

ELIGIBILITY:
Inclusion Criteria:

* Stage IA2-II non-small cell cancer patients who after complete resection.
* Two-round MRD tests confirm landmark undetectable MRD
* Expected survival ≥24 months
* ECOG PS 0-1
* Willing to accept MRD monitoring every 3 months for a total of 2 years after surgery

Exclusion Criteria:

* Patients who had previously undergone radiotherapy or chemotherapy or any other anti-tumor therapy
* Patients with a history of other malignancies in the past 5 years
* Any unstable systemic disease (eg, active infection, high-risk hypertension, unstable angina, congestive heart failure, etc.) or other conditions that investigators considered would limit the ability of the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Two-years disease free survival rates | 2 years
  The 2-year DFS rate of patients in both arms

SECONDARY OUTCOMES:
Use of adjuvant therapy | 2 years
  Differences in adjuvant therapy use between the Adaptive Therapy group (no adjuvant therapy if MRD persistently negative and initiation of adjuvant therapy if MRD positive) and the Standard Treatment Group
Questionnaire on Quality of Life | 2 years
  Differences in the Quality of Life between the Adaptive Therapy group (no adjuvant therapy if MRD persistently negative and initiation of adjuvant therapy if MRD positive) and the Standard Treatment Group, by using Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), and European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30, V3)
Five-years disease free survival rates | 5 years
  The 5-year DFS rate of patients in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Ma, M.D., Principal Investigator — Peking University Cancer Hospital & Institute, Beijing 100142, China
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No